CLINICAL TRIAL: NCT02289391
Title: Effect of Dexmedetomidine on Levels of Plasma Inflammatory Factor in Asthma Patients Undergoing General Anesthesia-single Center,Randomized,Double-blind，Controlled Trial
Brief Title: Effect of Dexmedetomidine on Levels of Plasma Inflammatory Factor in Asthma Patients Undergoing General Anesthesia
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Second Affiliated Hospital of Xi'an Jiaotong University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: Dexmedetomidine-14115
Record Dates: First submitted 2014-11-10; First posted 2014-11-13 (Estimated); Last update posted 2014-11-13 (Estimated); Status verified 2014-11

CONDITIONS: Anesthesia; Asthma
Keywords: Dexmedetomidine; Inflammatory factor; Inflammatory mediator; Cytokines; Asthma
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- non-asthma group (Placebo Comparator): * Non-asthma history
  * Infusion of normal saline(1μg/kg) at 10 minutes before anesthesia induction.
  * Infusion of normal saline at 0.4μg•kg-1•h-1during anesthesia maintenance.
  * Stop infusion of normal saline at 10 minutes before the end of surgery.
  Interventions: Drug: Anesthesia induction; Drug: Anesthesia maintenance
- Dexmedetomidine A (Experimental): * With a history of asthma
  * Infusion of dexmedetomidine(1μg/kg) at 10 minutes before anesthesia induction.
  * Infusion of dexmedetomidine at 0.4μg•kg-1•h-1during anesthesia maintenance.
  * Stop infusion of dexmedetomidine at 10 minutes before the end of surgery.
  Interventions: Drug: Anesthesia induction; Drug: Anesthesia maintenance; Drug: Assisted anesthesia
- Dexmedetomidine B (Experimental): * With a history of asthma
  * Infusion of dexmedetomidine(1μg/kg) at 10 minutes before anesthesia induction.
  * Infusion of dexmedetomidine at 0.7μg•kg-1•h-1during anesthesia maintenance.
  * Stop infusion of dexmedetomidine at 10 minutes before the end of surgery.
  Interventions: Drug: Anesthesia induction; Drug: Anesthesia maintenance; Drug: Assisted anesthesia
- Control group (Placebo Comparator): * With a history of asthma
  * Infusion of normal saline(1μg/kg) at 10 minutes before anesthesia induction.
  * Infusion of normal saline at 0.4μg•kg-1•h-1during anesthesia maintenance.
  * Stop infusion of normal saline at 10 minutes before the end of surgery.
  Interventions: Drug: Anesthesia induction; Drug: Anesthesia maintenance

INTERVENTIONS:
Drug: Anesthesia induction — -Intravenous injection midazolam 0.05 mg/Kg,fentanyl 4μg/Kg,etomidate 0.2 mg/Kg,cisatracurium 0.15 mg/Kg in proper order.
Drug: Anesthesia maintenance — * Continuous intravenous remifentanil O.2μg/(kg•h) and propofol 3~8mg/(kg•h).
  * Intermittent intravenous atracurium 0.05mg/kg. Maintain partial pressure of carbon dioxide(PETCO2) to 30~40 mmHg and bispectral index (BIS) to 45~60.
Drug: Assisted anesthesia — Intervention 'Assisted anesthesia' has been included in Arm Descriptions.
  Arms: Dexmedetomidine A; Dexmedetomidine B

SUMMARY:
The study try to illustrate the possible mechanisms of tending to induce airway spasms and the impact of dexmedetomidine on inflammatory reaction in general anesthesia patients with asthma，by detecting the differences of plasma inflammatory factor interleukin(IL)-4, IL-5, IL-13, IL-17, IL-33, MBP and immunoglobulin E(IgE) levels between asthma patients and non-asthma patients.

ELIGIBILITY:
Inclusion Criteria:

* Obtain informed consent
* Elective general anesthesia surgery, surgery time 1 ~ 3 hours.
* 20 patients with a history of asthma.
* 60 patients with no history of asthma.
* American Society of Anesthesiologists (ASA)classification:class I~II.
* Aged between 18 and 65 years old.

Exclusion Criteria:

* SBP≥180 mmHg or <90 mmHg, DBP≥110 mmHg or <60 mmHg.
* Serious heart, brain, liver, kidney, lung, endocrine diseases or serious infections.
* Hematopoietic dysfunction or bleeding tendency and hemorrhagic disease.
* A neuromuscular system disease.
* Airway and lung surgery.
* Predict possible or happened difficult airway.
* Immune function defect.
* Sure/suspected abuse of narcotic analgesics or drugs or alcohol dependence.
* The test drug allergy or have other contraindications in patients.
* Childbearing age women not to take appropriate contraception, pregnancy or lactation.
* Participated in other clinical drug research in the last 30 days.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2014-12; Primary Completion 2015-12 (Estimated); Study Completion 2015-12 (Estimated)

PRIMARY OUTCOMES:
IL-4，IL-5，IL-13, IL-17, IL-33 concentration in the Plasma | enter the operation room(T0)、10min after intubation(T1)、 skin incision(T2)、the end of surgery(T3)、24H after surgery(T4)
Histamine concentration | enter the operation room(T0)、10min after intubation(T1)、 skin incision(T2)、the end of surgery(T3)、24H after surgery(T4)
Myelin Basic Protein concentration （MBP) | enter the operation room(T0)、10min after intubation(T1)、 skin incision(T2)、the end of surgery(T3)、24H after surgery(T4)
IgE concentration | enter the operation room(T0)、10min after intubation(T1)、 skin incision(T2)、the end of surgery(T3)、24H after surgery(T4)

SECONDARY OUTCOMES:
Mean arterial pressure（MAP） | enter the operation room(T0)、10min after intubation(T1)、 skin incision(T2)、the end of surgery(T3)、24H after surgery(T4)
Heart rate（HR） | enter the operation room(T0)、10min after intubation(T1)、 skin incision(T2)、the end of surgery(T3)、24H after surgery(T4)
Respiratory rate（RR） | enter the operation room(T0)、10min after intubation(T1)、 skin incision(T2)、the end of surgery(T3)、24H after surgery(T4)

CONTACTS AND LOCATIONS:
Overall Officials: NIU XIAOLI, Principal Investigator — The second affiliated hospital of xi 'an jiaotong university

REFERENCES:
- [Background] Barnes PJ. The cytokine network in asthma and chronic obstructive pulmonary disease. J Clin Invest. 2008 Nov;118(11):3546-56. doi: 10.1172/JCI36130. PMID 18982161
- [Background] Saito A, Okazaki H, Sugawara I, Yamamoto K, Takizawa H. Potential action of IL-4 and IL-13 as fibrogenic factors on lung fibroblasts in vitro. Int Arch Allergy Immunol. 2003 Oct;132(2):168-76. doi: 10.1159/000073718. PMID 14600429
- [Background] Wen FQ, Kohyama T, Liu X, Zhu YK, Wang H, Kim HJ, Kobayashi T, Abe S, Spurzem JR, Rennard SI. Interleukin-4- and interleukin-13-enhanced transforming growth factor-beta2 production in cultured human bronchial epithelial cells is attenuated by interferon-gamma. Am J Respir Cell Mol Biol. 2002 Apr;26(4):484-90. doi: 10.1165/ajrcmb.26.4.4784. PMID 11919085
- [Background] Laporte JC, Moore PE, Baraldo S, Jouvin MH, Church TL, Schwartzman IN, Panettieri RA Jr, Kinet JP, Shore SA. Direct effects of interleukin-13 on signaling pathways for physiological responses in cultured human airway smooth muscle cells. Am J Respir Crit Care Med. 2001 Jul 1;164(1):141-8. doi: 10.1164/ajrccm.164.1.2008060. PMID 11435252
- [Background] Taniguchi T, Kidani Y, Kanakura H, Takemoto Y, Yamamoto K. Effects of dexmedetomidine on mortality rate and inflammatory responses to endotoxin-induced shock in rats. Crit Care Med. 2004 Jun;32(6):1322-6. doi: 10.1097/01.ccm.0000128579.84228.2a. PMID 15187514
- [Background] Kumar RK, Herbert C, Yang M, Koskinen AM, McKenzie AN, Foster PS. Role of interleukin-13 in eosinophil accumulation and airway remodelling in a mouse model of chronic asthma. Clin Exp Allergy. 2002 Jul;32(7):1104-11. doi: 10.1046/j.1365-2222.2002.01420.x. PMID 12100061